CLINICAL TRIAL: NCT05692622
Title: Exploring Effectiveness, Feasibility, and Acceptability of a Novel Home-based Complex Intervention for Children With Ataxia Telangiectasia: a Pilot Randomised Controlled Trial
Brief Title: Home-based Complex Intervention for Children With Ataxia Telangiectasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Munira Khan, Principal Investigator, University of Plymouth
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 3756
Record Dates: First submitted 2022-12-22; First posted 2023-01-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Ataxia Telangiectasia in Children; Ataxia Telangiectasia
Keywords: ataxia telangiectasia; ataxia; children; physical therapy; physiotherapy; exercise; yoga; breathing exercise; pilot RCT; complex intervention; home-based intervention
MeSH Terms: conditions — Ataxia Telangiectasia; Ataxia; Motor Activity | interventions — Yoga; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: A delayed start design will be used in this study
Who Masked: Outcomes Assessor
Masking Description: The participants will not be blinded to group allocation as both the groups will receive the same intervention, just at different time points. The principal investigator will not be blinded to the group allocation either as they will be the lead contact with the participants, monitoring their progress and engagement. The physiotherapist who will be carrying out outcome assessments will be blinded to the group allocation and not be made aware of the different timelines and structure of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early start group (Experimental): Participants in this group will receive a baseline monitoring period of 1 week, an active remotely supervised and monitored intervention period of 8 weeks and then an unsupervised but monitored follow up period of 4 months. They will be assessed at baseline (T0) and after one week (T1) to determine the sensitivity of the measures. They will then begin their intervention (T2) for a period of 8 weeks. At the end of the intervention phase (T3), assessment will be repeated that will also mark the beginning of a 16 weeks follow up period (T4), during this time they will have the choice to continue the exercises or stop them. At the end of the follow up period, assessment will be carried out again to measure any carry over effects.
  Interventions: Other: Whole-body exercise and respiratory exercise
- Delayed start group (Experimental): Participants in this group will receive a baseline monitoring period of 1 week, a control period of 8 weeks, an active remotely supervised and monitored intervention period of 8 weeks and then an unsupervised but monitored follow up period of 2 months. They will be assessed at baseline (T0) and after one week (T1) to determine the sensitivity of the measures. While the early start group receives their 8-week intervention, this group will not receive any intervention during this control period. At the end of 8 weeks, an assessment will be carried out for this group as well (T2). The participants will then begin their intervention (T3) for a period of 8 weeks. At the end of the intervention phase (T4), assessment will be repeated that will mark the beginning of an 8 weeks follow up period (T5), during this time they will have the choice to continue the exercises or stop them. At the end of the follow up period (T6), assessment will be carried out again to measure any carry over effects.
  Interventions: Other: Whole-body exercise and respiratory exercise

INTERVENTIONS:
Other: Whole-body exercise and respiratory exercise — The study involves an 8-week intervention involving whole-body and respiratory exercises. The whole-body exercise component will involve doing exercises while watching a total of 32 Comic Kids yoga movies. These movies have been adapted to suit the needs and abilities of the target population. For the first 7 weeks of intervention, children will be provided with 4 yoga movies for each week, providing around 67 minutes of exercise in each week. In the last week of intervention, children will have the choice to practice any 4 exercises of their choice from the 28 movies. The respiratory exercise component will involve watching a 10-minute-long movie that involves practicing different styles of breathing and breath holding. Participants will be provided a respiratory trainer to use while practicing these breathing exercises. Children will be asked to practice these breathing exercises by watching the movie at least 2 days each week.
  Other Names: Yoga and breathing exercises

SUMMARY:
Ataxia telangiectasia is a rare, genetic and progressive condition with no known cure. Therapies present a mainstream management option and have the potential to offer optimisation of fitness and general health. This pilot RCT aims to explore the effectiveness, feasibility, and acceptability of a co-produced home-based complex exercise intervention for children with ataxia telangiectasia. The study was designed through broad consultation with a collaborative of children and young people with A-T including family members, therapists, clinicians and researchers, called the A-Team collaborative (https://osf.io/edzn3/)

DETAILED DESCRIPTION:
Ataxia telangiectasia (A-T) usually presents in early childhood, primarily affecting the pulmonary, neurological and immunological systems. World-wide prevalence estimates vary between 1 in 40,000 and 1 in 100,000 live births. A-T typically presents with cerebellar ataxia in early childhood, generally before the age of four years, such that by early teenage most patients require a wheelchair for mobility. Oculomotor, extrapyramidal and peripheral nervous system problems occur in later childhood and adolescence. Lung disease and difficulties with feeding, swallowing and nutrition are also common. A-T also carries a high risk of malignancy, and life-expectancy for individuals with A-T is decreased, with survival time of 25 years.

People living with A-T require coordinated multi-disciplinary care to optimally manage their complex needs. Symptomatic management and rehabilitation is advocated to improve quality of life and minimize complications that could increase morbidity and mortality. However, the feasibility and acceptability of allied health interventions and outcome measures for this population group are under-researched. Parents participating in a research engagement meeting reported being unclear about how best to deal with the signs and symptoms of A-T at home, how to find help and how and when to access support. This uncertainty is echoed by therapists treating children and adults with ataxia. Evidence is lacking about what type of therapy is needed and how it might be best delivered. The investigators intend to address these concerns and perspectives by investigating the effectiveness, feasibility, and acceptability of a home-based exercise intervention that offers therapeutic interventions for the impairments, activity limitations, and participation restrictions related to A-T.

An extensive review undertaken at the beginning of this overall project scoping the evidence on care and management of A-T provided by allied health professionals and nurses, identified a range of interventions that reportedly positively impact A-T related impairments, together with quality of life, indicating that outcomes can be improved for this population. Through i) considerable and robust engagement to date with key stakeholders (including parents, older children and young adults with A-T, physiotherapists, occupational therapists and charity workers), and ii) evidence from other research studies involving pediatric populations with the same or similar health conditions which indicate the potential benefits of yoga and breathing exercises in optimizing health, fitness and wellbeing, the investigators have identified a strong need for this study.

Objectives

1. Assess the effectiveness of the complex home-based exercise intervention on physical function, respiratory muscle strength, participation, and quality of life
2. Investigate the feasibility of the complex home-based exercise intervention in terms of:

   1. online and remote delivery by a multi-disciplinary health profession team with an allied health-professional lead (exploring factors such as undertaking online assessment, supervising exercise and wider trial activities, supporting participants and their families and monitoring safety)
   2. participant and families' abilities to undertake the exercises (exploring factors such as frequency and duration of exercises, and length of the intervention programme)
   3. use of a digital platform for accessing exercise movies and sharing feedback and experience with research team and other participating families
3. Investigate the feasibility of the home-based clinical trial design in terms of:

   1. participant recruitment and online consent taking
   2. online and remote delivery of home-based intervention
   3. online assessments at four different time points and engagement with extensive trial-based battery of outcome measures
   4. conducting exit interviews online
   5. use of the digital platform for trial involvement
4. Determine intervention fidelity in terms of:

   1. the degree to which the intervention is implemented as intended
   2. frequency, intensity and duration of exercise interventions
   3. what were the barriers faced (if any) and how were they addressed?
   4. what were the facilitators (if any) for undertaking the exercises?
5. Explore the perception and experiences of parents/legal guardians and children with A-T undertaking the exercises regarding engagement, effectiveness, and acceptability of the intervention
6. Analyse the data of this pilot study to

   1. Select the most appropriate outcome measure and inform design of an onward RCT
   2. Make recommendations about whether a fully powered trial may be undertaken depending on whether the feasibility of the home-based exercise intervention and the home-based clinical trial design is established.
   3. Inform the power calculation for the subsequent RCT using the outcome data from this study

The project that this study is a part of, is funded by Action for A-T and supported for PPIE and recruitment by the A-T Society. Dr Lisa Bunn is the principal investigator and Dr Tracey Parkin the co-principal investigator of this project. A list of all the collaborators of this project is available on the following link- https://osf.io/edzn3/

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of A-T confirmed clinically
* Aged 4-11 years
* Able to walk independently (with no or only intermittent support) over 10 metres and stand unaided for 1 minute
* Able to communicate in English either independently or with the assistance of their parent/legal guardian (where parent/guardian is able to communicate in English) or using a translator arranged by the participating family
* Has the ability to assent and parents/legal guardians have the ability to give consent on their child's behalf

Exclusion Criteria:

* Those with other/additional diagnoses thought by the study team to probably compromise the intervention, e.g. with significant intellectual disability
* Currently undergoing cancer therapies or acutely unwell
* Children who are participants of another trial/intervention programme
* Non-UK based families

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Scale for the Assessment and Rating of Ataxia; to assess change in score between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  Scale for the Assessment and Rating of Ataxia (SARA) is a reliable and valid clinical scale used to measure the severity of ataxia. It has eight categories with accumulative score ranging from 0 (no ataxia) to 40 (most severe ataxia); where higher score indicates worse outcomes. SARA was selected as the primary outcome measure as it is a validated tool that is widely used in paediatric population. It has also been successfully used in A-T population in the context of clinical trials of intervention and is validated for remote assessment.

SECONDARY OUTCOMES:
Spirometry to measure slow vital capacity; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  A spirometer (MIR Spirobank smart spirometer) will be used to measure the respiratory muscle strength. It measures lung function, specifically the volume of air inspired and expired by the lungs. The investigators will use this test to measure slow vital capacity (SVC). SVC is the volume of air expired, through an unforced maneuver; where higher score indicates better outcomes
Spirometry to measure forced vital capacity; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  A spirometer (MIR Spirobank smart spirometer) will be used to measure the respiratory muscle strength. It measures lung function, specifically the volume of air inspired and expired by the lungs. The investigators will use this test to measure forced vital capacity (FVC). FVC is the maximum amount of air that can be forcibly exhaled from lungs after fully inhaling; where higher score indicates better outcomes.
Spirometry to measure forced expiratory volume in the first second; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  A spirometer (MIR Spirobank smart spirometer) will be used to measure the respiratory muscle strength. It measures lung function, specifically the volume of air inspired and expired by the lungs. The investigators will use this test to measure forced expiratory volume in the first second (FEV1). FEV1 is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration; where higher score indicates better outcomes.
Spirometry to measure peak expiratory flow; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  A spirometer (MIR Spirobank smart spirometer) will be used to measure the respiratory muscle strength. It measures lung function, specifically the volume of air inspired and expired by the lungs. The investigators will use this test to measure peak expiratory flow (PEF). PEF is the volume of air forcefully expelled from the lungs in one quick exhalation; where higher score indicates better outcomes.
Pediatric Evaluation of Disability Inventory Computer Adaptive Test; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) measures abilities in the domains of daily activities, mobility, social/cognitive, and responsibility. The domains of daily activities, mobility, and social/cognitive are rated on a 4 point difficulty scale with responses ranging from 'Unable' to 'Easy'; where higher score indicates better outcomes. The responsibility domain is rated on a 5 point scale with responses ranging from 'Adult/caregiver has full responsibility; the child does not take any responsibility' to 'Child takes full responsibility without any direction, supervision or guidance from an adult/caregiver'; where higher score indicates better outcomes.
EuroQuol-5Dimensions-Youth scale; to assess change in scores between different time points | Early start group assessments at baseline, week 1, week 9, and week 25; delayed start group assessments at baseline, week 1, week 9, week 17,and week 25
  EuroQuol-5Dimensions-Youth (EQ-5D-Y) measures quality of life in the following dimensions of health: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems, and extreme problems; based on the response, scores are assigned between 1 to 3, where higher score indicates worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Plymouth, Plymouth, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The investigators are exploring an intervention on a group of people with a rare condition which is unlikely to ever be fully powered owing to the small population size. Presentation of anonymised raw effectiveness data will therefore be made available with publications in order for future research to build on these results on an international scale should this opportunity arise.
Supporting Information: Study Protocol, SAP
Time Frame: Anticipated in 2024
Access Criteria: Anonymised IPD will not be shared until the study is published and available in public domain. It is anticipated to be shared as supplementary data if not embedded within the report.
URL: https://osf.io/edzn3/

REFERENCES:
- [Background] Rothblum-Oviatt C, Wright J, Lefton-Greif MA, McGrath-Morrow SA, Crawford TO, Lederman HM. Ataxia telangiectasia: a review. Orphanet J Rare Dis. 2016 Nov 25;11(1):159. doi: 10.1186/s13023-016-0543-7. PMID 27884168
- [Background] van Os NJH, Haaxma CA, van der Flier M, Merkus PJFM, van Deuren M, de Groot IJM, Loeffen J, van de Warrenburg BPC, Willemsen MAAP; A-T Study Group. Ataxia-telangiectasia: recommendations for multidisciplinary treatment. Dev Med Child Neurol. 2017 Jul;59(7):680-689. doi: 10.1111/dmcn.13424. Epub 2017 Mar 20. PMID 28318010
- [Background] Taylor et al. Ataxia-telangiectasia in children Guidance on diagnosis and clinical care. Ataxia-Telangiectasia Society. 2014; 1-31
- [Background] McGrath-Morrow SA, Gower WA, Rothblum-Oviatt C, Brody AS, Langston C, Fan LL, Lefton-Greif MA, Crawford TO, Troche M, Sandlund JT, Auwaerter PG, Easley B, Loughlin GM, Carroll JL, Lederman HM. Evaluation and management of pulmonary disease in ataxia-telangiectasia. Pediatr Pulmonol. 2010 Sep;45(9):847-59. doi: 10.1002/ppul.21277. PMID 20583220
- [Background] Reiman A, Srinivasan V, Barone G, Last JI, Wootton LL, Davies EG, Verhagen MM, Willemsen MA, Weemaes CM, Byrd PJ, Izatt L, Easton DF, Thompson DJ, Taylor AM. Lymphoid tumours and breast cancer in ataxia telangiectasia; substantial protective effect of residual ATM kinase activity against childhood tumours. Br J Cancer. 2011 Aug 9;105(4):586-91. doi: 10.1038/bjc.2011.266. Epub 2011 Jul 26. PMID 21792198
- [Background] Amirifar P, Ranjouri MR, Yazdani R, Abolhassani H, Aghamohammadi A. Ataxia-telangiectasia: A review of clinical features and molecular pathology. Pediatr Allergy Immunol. 2019 May;30(3):277-288. doi: 10.1111/pai.13020. Epub 2019 Mar 20. PMID 30685876
- [Background] Perlman SL, Boder Deceased E, Sedgewick RP, Gatti RA. Ataxia-telangiectasia. Handb Clin Neurol. 2012;103:307-32. doi: 10.1016/B978-0-444-51892-7.00019-X. No abstract available. PMID 21827897
- [Background] Hartley H, Carter B, Bunn L, Pizer B, Lane S, Kumar R, Cassidy E. E-Survey of Current International Physiotherapy Practice for Children with Ataxia Following Surgical Resection of Posterior Fossa Tumour. J Rehabil Med Clin Commun. 2019 Dec 30;2:1000020. doi: 10.2340/20030711-1000020. eCollection 2019. PMID 33884121
- [Background] Cassidy E, Reynolds F, Naylor S, De Souza L. Using interpretative phenomenological analysis to inform physiotherapy practice: an introduction with reference to the lived experience of cerebellar ataxia. Physiother Theory Pract. 2011 May;27(4):263-77. doi: 10.3109/09593985.2010.488278. Epub 2010 Aug 26. PMID 20795878
- [Background] Ross LJ, Capra S, Baguley B, Sinclair K, Munro K, Lewindon P, Lavin M. Nutritional status of patients with ataxia-telangiectasia: A case for early and ongoing nutrition support and intervention. J Paediatr Child Health. 2015 Aug;51(8):802-7. doi: 10.1111/jpc.12828. Epub 2015 Feb 6. PMID 25656498
- [Background] Galantino ML, Galbavy R, Quinn L. Therapeutic effects of yoga for children: a systematic review of the literature. Pediatr Phys Ther. 2008 Spring;20(1):66-80. doi: 10.1097/PEP.0b013e31815f1208. PMID 18300936
- [Background] Felix E, Gimenes AC, Costa-Carvalho BT. Effects of inspiratory muscle training on lung volumes, respiratory muscle strength, and quality of life in patients with ataxia telangiectasia. Pediatr Pulmonol. 2014 Mar;49(3):238-44. doi: 10.1002/ppul.22828. Epub 2013 Aug 19. PMID 23956159
- [Background] Kepenek-Varol B, Gurses HN, Icagasioglu DF. Effects of Inspiratory Muscle and Balance Training in Children with Hemiplegic Cerebral Palsy: A Randomized Controlled Trial. Dev Neurorehabil. 2022 Jan;25(1):1-9. doi: 10.1080/17518423.2021.1905727. Epub 2021 Apr 1. PMID 33792496
- [Background] Nissenkorn A, Borgohain R, Micheli R, Leuzzi V, Hegde AU, Mridula KR, Molinaro A, D'Agnano D, Yareeda S, Ben-Zeev B. Development of global rating instruments for pediatric patients with ataxia telangiectasia. Eur J Paediatr Neurol. 2016 Jan;20(1):140-6. doi: 10.1016/j.ejpn.2015.09.002. Epub 2015 Sep 25. PMID 26493850
- [Background] Broccoletti T, Del Giudice E, Cirillo E, Vigliano I, Giardino G, Ginocchio VM, Bruscoli S, Riccardi C, Pignata C. Efficacy of very-low-dose betamethasone on neurological symptoms in ataxia-telangiectasia. Eur J Neurol. 2011 Apr;18(4):564-70. doi: 10.1111/j.1468-1331.2010.03203.x. Epub 2010 Sep 14. PMID 20840352
- [Background] Russo I, Cosentino C, Del Giudice E, Broccoletti T, Amorosi S, Cirillo E, Aloj G, Fusco A, Costanzo V, Pignata C. In ataxia-teleangiectasia betamethasone response is inversely correlated to cerebellar atrophy and directly to antioxidative capacity. Eur J Neurol. 2009 Jun;16(6):755-9. doi: 10.1111/j.1468-1331.2009.02600.x. PMID 19475758
- [Background] Tai G, Corben LA, Woodcock IR, Yiu EM, Delatycki MB. Determining the Validity of Conducting Rating Scales in Friedreich Ataxia through Video. Mov Disord Clin Pract. 2021 Apr 6;8(5):688-693. doi: 10.1002/mdc3.13204. eCollection 2021 Jul. PMID 34307740